CLINICAL TRIAL: NCT00882258
Title: A Phase II, Multicenter, Randomized, Placebo-controlled, Double-blinded Study of the Selective Progesterone Receptor Modulator Proellex (CDB-4124) in Pre-menopausal Women With Symptomatic Leiomyomata
Brief Title: Study of Proellex in Pre-menopausal Women With Symptomatic Uterine Fibroids
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ZPU-003
Record Dates: First submitted 2009-04-14; First posted 2009-04-16 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Uterine Fibroids
Keywords: Uterine fibroids
MeSH Terms: conditions — Leiomyoma | interventions — telapristone acetate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 12.5 mg Proellex (Experimental): Proellex 12.5 mg daily
  Interventions: Drug: 12.5 mg Proellex
- 25 mg Proellex daily (Experimental): Proellex 25 mg
  Interventions: Drug: 25 mg Proellex
- Placebo (Placebo Comparator): Placebo daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 12.5 mg Proellex — 12.5 mg Proellex administered orally daily
  Other Names: CDB-4124; Telapristone acetate
  Arms: 12.5 mg Proellex
Drug: 25 mg Proellex — 25 mg Proellex administered orally daily
  Other Names: CDB-4124; Telapristone acetate
  Arms: 25 mg Proellex daily
Drug: Placebo — Administered orally daily
  Other Names: Dummy
  Arms: Placebo

SUMMARY:
Two (2) dose levels of Proellex or placebo will be administered once-daily for up to 91 days. Following screening and a pre-treatment endometrial biopsy, subjects will be followed monthly for the three month treatment phase.

DETAILED DESCRIPTION:
Two (2) dose levels of Proellex or placebo will be administered once-daily for up to 91 days. Following screening and a pre-treatment endometrial biopsy, subjects will be followed monthly for the three month treatment phase. At the three-month treatment visit, subjects will be entered into an open-label extension treatment protocol, if deemed eligible. At four months after their first treatment visit, subjects not electing to enter the open-label study will be assessed at a final follow-up visit.

ELIGIBILITY:
Inclusion Criteria:

* At least one leiomyoma must have been identifiable and measurable by abdominal/pelvic ultrasound.
* Must have had a history of one or both of the following leiomyomata-associated symptoms, excessive menstrual bleeding, or pain

Exclusion Criteria:

* Post-menopausal women, as defined as one or more of the following:

  1. six months or more (immediately prior to Screening visit) without a menstrual period, or
  2. prior hysterectomy and/or oophorectomy
* Subjects with documented endometriosis

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 144 (Actual)
Dates: Start 2006-03; Primary Completion 2007-03 (Actual); Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
To evaluate Proellex administered once daily in pre-menopausal women with symptomatic leiomyomata | 91 days

SECONDARY OUTCOMES:
To evaluate the efficacy of two different doses of Proellex versus placebo for the treatment of symptomatic leiomyomata | 91 days

CONTACTS AND LOCATIONS:
Overall Officials: Andre VanAs, PhD, MD, Study Director — Repros Therapeutics Inc.
Locations (16):
- United States (16):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - Women's Health Research, Phoenix, Arizona
  - Arizona Wellness Centre for Women, Phoenix, Arizona
  - Visions Clinical Research Tuscon, Tuscon, Arizona
  - Medical Centre for Clinical Research, San Diego, California
  - Women's Health Care, Inc., San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Visions Clinical Research, Boynton Beach, Florida
  - Miami Research Associates, Women's Health Studies, Miami, Florida
  - Insignia Clinical Research (Tampa Bay Women's Center), Tampa, Florida
  - Caring for Women, Las Vegas, Nevada
  - Affiliated Clinical Research, Inc., Las Vegas, Nevada
  - SC Clinical Research Center, Columbia, South Carolina
  - Advances in Health Inc., Houston, Texas
  - Obstetrical & Gynecolgical Associates, PA (OGA), Houston, Texas
  - Women's Clinical Research Centre, Seattle, Washington